CLINICAL TRIAL: NCT07164911
Title: Prédiction Des réponses du Patient Porteur d'Une Insuffisance Cardiaque à Fraction d'éjection altérée à Une Phase II de réadaptation Cardiaque
Brief Title: Predictive Factors of Response to Phase II Cardiac Rehabilitation in Heart Failure With Reduced Ejection Fraction
Acronym: PrédicRéa
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Corbie (Other Government)
Responsible Party: Sponsor
Other Study IDs: Centre hospitalier de Corbie; 2025-A01575-44 (Other: Agence Nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2025-08-24; First posted 2025-09-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: HFrEF - Heart Failure With Reduced Ejection Fraction; Cardiac Rehabilitation; Exercise Training; Exercise Adaptations; Exercise Intolerance; Exercise Intervention
Keywords: Exercise-based cardiac rehabilitation in patients with reduced left ventricular ejection fraction; VO2peak; MicroRNA; Muscle Oxygenation; arterial stiffness; cardiac output; stroke volume; Oxygen alveolar-arterial gradient; alveolar ventilation; minute ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Exercise intolerance, measured as peak oxygen consumption (VO₂peak) during exercise in patients with heart failure with reduced ejection fraction (HFrEF). Change in VO₂peak (ΔVO₂peak), which serves as a prognostic marker for HFrEF engaged in exercise based cardiac rehabilitation program (ExCR). Responders to ExCR generally show improved cardiac function but some patients with HFrEF do not respond to ExCR. VO₂peak depends on three major components of oxygen transport: Pulmonary (lungs), circulatory (heart and vessels) and skeletal muscle (oxygen utilization) functions. These physiological responses to ExCR may be influenced by epigenetic regulation, specifically the expression of circulating microRNAs (c-miRNAs).

Linking non-invasive measurements and epigenetic markers could 1) identify which component of the oxygen transport chain is most impaired and 2) allow personalized interventions to maximize VO₂peak improvements.

The primary objective of this stidy is to assess the association between changes in VO₂peak during exercise training and circulating microRNA expression (miR-146a, miR-191, miR-23a, miR-140, miR-1, miR-21, miR-133a, miR-17-5p, miR-3200-3p).

The secondary objective is to examine the relationship between pulmonary, cardiovascular, and neuromuscular adaptations to exercise and circulating microRNA expression.

DETAILED DESCRIPTION:
Key Takeaways VO₂peak is a clinically relevant, prognostic measure in HFrEF. .ExCR benefits are heterogeneous, partly due to variable cardiac and muscular adaptations. c-miRNAs may mediate or indicate the molecular response to ExCR. c-miRNAs may Enhance pulmonary, cardiac, or muscular adaptations → improved VO₂peak, or, if maladaptive, contribute to fatigue → explaining non-response.

Goal Connect ΔVO₂peak with cellular precursors of adaptation, providing a mechanistic understanding of CR responses.

Method 62 patients with HFrEF will be engaged in a this prospective, single-center cohort follow-up study with a prognostic aim and minimal risk to human participants.

Peak values of oxygen uptake, cardiac hemodynamics, cerebral and muscle oxygenation, non-coding RNA will be measured before and after Exercise based cardiac rehabilitation during a cardiopulmonary exercise testing. All the patients will perform a force - velocity test in order to prescribe an individualized resistance training program.

Originality of study: Combines non-invasive physiological measurements during exercise and biomarker (c-miRNA) analysis before and after ExCR.

Scientific and Clinical Significance

Linking non-invasive measurements and epigenetic markers could:

1. Identify which component of the oxygen transport chain is most impaired.
2. Combining physiological and molecular assessments could guide tailored rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with reduced ejection fraction < 40%
* NYHA functional class ≥ II
* Clinically stable for at least 6 weeks
* On optimized medical therapy for at least 6 weeks
* Prescription for phase II cardiac rehabilitation
* BMI between 20-30 kg·m-²
* Physical activity level: sedentary or physically active but untrained
* Signed informed consent to participate in the study
* Affiliation to the French national health insurance system

Exclusion Criteria:

* Contraindication to regular adapted physical activity
* Uncontrolled arterial hypertension
* Secondary respiratory disease such as emphysema or chronic obstructive pulmonary disease (COPD)
* Secondary cardiovascular disease
* Individuals under legal protection or deprived of liberty
* Pregnant or breastfeeding women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patient with altered left ventricular ejection fraction
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
ΔVO₂peak | Day 1 : baseline value of peak oxygen consumption (preVO₂peak) Day 21: post value of peak oxygen consumption (post VO₂peak)
  Variation in peak oxygen consumption during exercise (ΔVO₂peak = postVO₂peak - preVO₂peak), expressed as the percentage change from baseline after exercise training.
circulating microRNAs | Day 1 : baseline expression of miRNAs (pre-miRNAs) Day 21: post values of miRNAs expression (post-miRNAs)
  Expression of circulating microRNAs (c-miRNAs): miR-146a, miR-191, miR-23a, miR-140, miR-1, miR-21, miR-133a, miR-17-5p, miR-3200-3p

SECONDARY OUTCOMES:
Changes in pulmonary ventilation | Day 1: pulmonary ventilation at baseline (preVE, L·min-¹) Day 21: post value of pulmonary ventilation (postVE, L·min-¹)
  Changes (pre-post exercise training) in pulmonary ventilation (VE, L·min-¹).
Changes in alveolar ventilation with exercise training | Day 1: alveolar ventilation at baseline (postVA, mL·min-¹) Day 21: post value of alveolar ventilation (postVA, mL·min-¹)
  Changes (pre-post exercise training) in alveolar ventilation (VA, mL·min-¹)
Changes in alveolar-arterial oxygen pressure difference with exercise training | Day 1: baseline alveolar-arterial oxygen pressure difference value (prePA-aO₂, mmHg) Day 21: post value of alveolar-arterial oxygen pressure difference (postPA-aO₂, mmHg)
  Changes (pre-post exercise training) in alveolar-arterial oxygen pressure difference (PA-aO₂, mmHg)
Changes in cardiac index with exercise training | Day 1: baseline value of cardiac index (preCI, L·min-¹·m-²) Day 21: post value of cardiac index (postCI, L·min-¹·m-²)
  Changes (pre-post exercise training) in cardiac index (CI, L·min-¹·m-²)
Changes in arterial stiffness with exercise training | Day 1: baseline value of arterial stiffness (prePWV, m·s-¹) Day 21: post value of arterial stiffness (postPWV, m·s-¹)
  Changes (pre-post exercise training) in arterial stiffness (PWV, m·s-¹)
Changes in muscle oxygen saturation | Day 1: baseline value of muscle oxygen saturation (preSmO₂, %) Day 2: post value of muscle oxygen saturation (postSmO₂, %)
  Changes (pre-post exercise training) in muscle oxygen saturation (SmO₂, %)
Changes in cerebral oxygen saturation with exercise training | Day 1: baseline value of cerebral oxygen saturation (%) Day 21: baseline value of cerebral oxygen saturation '%)
  Changes (pre-post exercise training) in cerebral oxygen saturation (%)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie Leprêtre, Professor, Study Director — Université de Rouen Normandie, UFR-STAPS; Francesco Orlando, MD, Principal Investigator — Centre Hospitalier de Corbie
Locations (1):
- Hospital center of Corbie, Corbie, France